CLINICAL TRIAL: NCT01912586
Title: A Non-randomised Controlled Trial of Early Intervention to Preserve Erectile Function After Laparoscopic Resection for Rectal Cancer
Brief Title: Early Intervention for Erectile Dysfunction After Laparoscopic Resection for Rectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Haijun Deng, MD, PhD, Associate professor, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NanFang2013035
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-02

CONDITIONS: Rectal Tumors; Erectile Dysfunction
Keywords: erectile dysfunction; laparoscopic surgery; rectal cancer; sildenafil; vacuum erection device
MeSH Terms: conditions — Rectal Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (No Intervention): Patients receive no interventions for ED after laparoscopic surgery
- Arm B (Experimental): sildenafil 25mg/day nightly without vacuum erection device for 3 months after surgery within one or two weeks.
  Interventions: Other: vacuum erection device
- Arm C (Experimental): sildenafil 25mg/day nightly and together with using vacuum erection device to make erections for 10-15 minutes/day for 3 months after surgery within one or two weeks.
  Interventions: Other: vacuum erection device

INTERVENTIONS:
Other: vacuum erection device — sildenafil: 25mg/day nightly for 3 months vacuum erection device: make erections for 10-15 minutes/day for 3 months
  Other Names: sildenafil
  Arms: Arm B; Arm C

SUMMARY:
Although the high prevalence of erectile dysfunction (ED) was detected among male patients after the treatment for colorectal cancer, published reports depicting the erectile dysfunction experience of patients with colorectal cancer ot underpin service development are insufficient. Furthermore,unlike patients with prostate cancer, men with colorectal cancer are not routinely offered information and treatment for erectile dysfunction.However, investigations on patients after surgery for prostate cancer could provide some potentially useful insights. The ability of sildenafil and vacuum erection device (VED) to aid in the return of erections after nerve-sparing radical prostatectomy has been established, which may benefit rectal cancer patients after surgery with ED.

Laparoscopic surgery, although technically demanding and associated with a long learning curve, has the advantage of clear visualization for the smallest structures,including the autonomic nerves. Laparoscopic resection for rectal cancer could thus facilitate preservation of the pelvic autonomic nerves.

This study aimed to identify whether early intervention is effective at reducing the rate of ED at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 < Age < 70
2. Sexually active men without the consistent use of erectile aids pre-operatively
3. Rectal cancer confirmed by histology
4. Undergoing a bilateral nerve sparing laparoscopic rectal resection
5. IIEF-5 domain score > =20 before surgery
6. Presence of a female sexual partner
7. Willingness to participate in clinical research as evidenced by their signature on the informed consent form

Exclusion Criteria:

1. Has a history of cardiac failure, angina, or life-threatening arrhythmia within the past 6 months
2. Has taken or has been prescribed nitrate medication in any form in the last 6 months
3. Contraindication to sildenafil (e.g. nitrates, hypersensitivity)
4. Contraindication to vacuum erection device (e.g. coagulation abnormality, stick cell disease)
5. Men with a history of known penile deformity or Peyronie's disease
6. Pre or postoperative androgen therapy

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in sexual function based on the (IIEF)-5 score and NPT | 3 months
  Summarized according to assigned treatment group. Erectile Dysfunction is defined by The International Index of Erectile Dysfunction(IIEF)-5 score and Nocturnal penile tumescence(NPT).
Changes in sexual function based on the (IIEF)-5 score and NPT | 6 months
  Summarized according to assigned treatment group. Erectile Dysfunction is defined by The International Index of Erectile Dysfunction(IIEF)-5 score and Nocturnal penile tumescence(NPT).
Changes in sexual function based on the (IIEF)-5 score and NPT | 12 months
  Summarized according to assigned treatment group. Erectile Dysfunction is defined by The International Index of Erectile Dysfunction(IIEF)-5 score and Nocturnal penile tumescence(NPT).

SECONDARY OUTCOMES:
Compliance and overall patient satisfaction based on the self reported compliance diary and IIEF-5 score and NPT | 12 months
  Summarized according to assigned treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Dowswell G, Ismail T, Greenfield S, Clifford S, Hancock B, Wilson S. Men's experience of erectile dysfunction after treatment for colorectal cancer: qualitative interview study. BMJ. 2011 Oct 18;343:d5824. doi: 10.1136/bmj.d5824. PMID 22010127
- [Background] McGlone ER, Khan O, Flashman K, Khan J, Parvaiz A. Urogenital function following laparoscopic and open rectal cancer resection: a comparative study. Surg Endosc. 2012 Sep;26(9):2559-65. doi: 10.1007/s00464-012-2232-5. Epub 2012 Apr 5. PMID 22476834
- [Background] Lange MM, van de Velde CJ. Urinary and sexual dysfunction after rectal cancer treatment. Nat Rev Urol. 2011 Jan;8(1):51-7. doi: 10.1038/nrurol.2010.206. Epub 2010 Dec 7. PMID 21135876